CLINICAL TRIAL: NCT03435432
Title: Investigating the Molecular Mechanisms Underpinning Glucose Stimulated Release of Stored Enteral Lipid in Humans
Brief Title: Plasma Lipid Response to Glucose Drink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Glucose Plasma 15-9025
Record Dates: First submitted 2018-02-09; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-01

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias | interventions — Glucose; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucose (Active Comparator): 50 grams of glucose in 50 ml water
  Interventions: Dietary Supplement: Glucose
- Water (Placebo Comparator): 50 ml water
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Glucose — Glucose drink
  Arms: Glucose
Dietary Supplement: Water — Control
  Arms: Water

SUMMARY:
During dietary fat absorption, the gut packages the majority of the fats into lipid particles that are secreted into blood circulation. The gut is also capable of storing a considerable amount of fats that can be released at a later time upon receiving certain stimulus signals. One of the signals is glucose ingestion. This protocol examines blood lipid responses to a glucose drink. Participants drink a fatty formula and 5 hours later drink either a glucose solution or water (as control), in one of two randomized study visits. Blood lipid levels are monitored throughout the study period.

DETAILED DESCRIPTION:
Participants are recruited after obtaining informed consent. They first have a high fat liquid formula. 5 hours later, they drink 50 grams of glucose in 50 ml of water in one visit and 50 ml of water in another. The 2 visits are randomized. Blood samples are taken before and after they drink the high fat liquid formula, and continued until 3 hours after they drink glucose or water. Lipid levels in the blood samples are measured in the lab.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 to 60 years requiring endoscopy and duodenal biopsies for clinical indications, with no contraindications to the procedure, as judged by Dr. Bookman.
* Body mass index 20 to 27 kg/m2

Exclusion Criteria:

* Patients with active inflammatory bowel disease
* Patients with Celiac disease, exocrine pancreatic insufficiency or small bowel malabsorption
* Patients with active bowel malignancy
* Patients with diabetes mellitus or known/ suspected motility disorders of the gut
* Patients with decompensated liver disease
* Patients on ezetemibe or bile acid sequestrants
* Unstable cardiac or respiratory disease
* Any changes to medication in the preceding month.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2016-06-16 (Actual); Study Completion 2016-06-16 (Actual)

PRIMARY OUTCOMES:
Blood lipid responses to glucose drink | 8 hours
  Blood lipid levels are measured after drinking a glucose solution

CONTACTS AND LOCATIONS:
Locations (1):
- Tornto General Hospital, UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No